CLINICAL TRIAL: NCT01207492
Title: A Multi-Center Single Agent Phase II Study of the Efficacy of Nilotinib in Patients With Relapsed or Metastatic Pigmented Villonodular Synovitis/Tenosynovial Giant Cell Tumor/Diffuse-Type Giant Cell Tumor
Brief Title: Nilotinib in Patients With Relapsed or Metastatic Pigmented Villonodular Synovitis/Tenosynovial Giant Cell Tumor/Diffuse-Type Giant Cell Tumor
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew J. Wagner, MD, PhD (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Andrew J. Wagner, MD, PhD, Sponsor, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-179; YUS23T (Other: Novartis)
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pigmented Villonodular Synovitis; Diffuse-type Giant Cell Tumor; Tenosynovial Giant Cell Tumor
Keywords: nilotinib
MeSH Terms: conditions — Synovitis, Pigmented Villonodular; Giant Cell Tumor of Tendon Sheath | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib (Experimental): Nilotinib 200 mg taken as 400 mg twice daily, continuously
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — Taken orally twice daily

SUMMARY:
Nilotinib is a drug that is used to treat a form of a blood cancer called leukemia. Nilotinib works by blocking the action of a protein that might be important for the growth of pigmented villonodular synovitis (PVNS). In this research study the investigators are testing whether nilotinib can stop the growth of PVNS or improve the symptoms experienced from PVNS.

DETAILED DESCRIPTION:
* In this research study, each cycle of study drug dosing will last 4 weeks (28 days). During each cycle, participants will take nilotinib by mouth twice daily. During the first cycle, participants will come to the clinic on Days 1 and 8. For Cycles 2-4 and every 3 cycles thereafter, they will come to the clinic on Day 1.
* The following tests and procedures will be performed at specific time points during study treatment: MRI or CT scans; physical examinations; vital signs; blood work; questionnaires and EKG.
* Participants may continue in this research study for as long as they do not have serious side effects or their disease does not get worse.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of recurrent PVNS ( or diffuse-type giant cell tumor or tenosynovial giant cell tumor) that is unresectable, metastatic, or for which the patient refuses surgical intervention
* Progressive disease in the last 12 months, as demonstrated by imaging or clinical appearance of new tumors, in the opinion of the treating investigator
* At least one site of measurable disease according to RECIST 1.1 on MRI (or CT scan for metastatic disease)
* Any number or type of prior systemic therapies, with the exception of known or suspected CSF1 receptor inhibitors as outlined in exclusion criteria below
* 18 years of age or older
* Life expectancy greater than 6 months
* ECOG Performance Status of 0, 1 or 2
* Normal organ and marrow function as defined in the protocol
* QTc less than or equal to 450 ms on 12-lead ECG
* Negative urine or serum pregnancy test within days of start of study drug administration for women of childbearing potential.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 3 months following study drug discontinuation

Exclusion Criteria:

* Prior treatment with known or suspected CSF1 receptor inhibitor, including nilotinib, imatinib, sunitinib, or sorafenib, or other approved or investigational tyrosine kinase inhibitors used for treatment of diffuse-type giant cell tumor
* Concurrent treatment with other investigational agents
* Inability to tolerate or contraindication to MRI scanning for participants with localized disease
* Impaired cardiac function
* Current treatment with strong CYP3A4 inhibitors that cannot either be discontinued or switched to a different medication prior to starting study drug
* Current treatment with any medications that have the potential to prolong the QT interval and that cannot either be discontinued or switched to a different medication prior to starting study drug
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug
* Acute or chronic pancreatic disease
* Acute or chronic liver disease
* Another primary malignant disease requiring systemic treatment or radiation
* History of significant congenital or acquired bleeding disorder unrelated to cancer
* Major surgery within 28 days prior to Day 1 of the study
* Treatment with other investigational agents within 28 days of day 1
* History of non-compliance to medical regimens or inability to grant consent
* Women who are pregnant or breastfeeding
* Other comorbidities that would interfere with study participation or safety in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Wagner, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UT MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nilotinib
Started | 17
Completed | 2
Not Completed | 15
Not completed — Still on study | 1
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 1
Not completed — Progressive disease | 3
Not completed — Toxicity | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.35 (13.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival
Description: To estimate progression free survival at 6 months in participants with recurrent PVNS treated with nilotinib. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants with PFS
Arm/Group | Nilotinib
Number analyzed (Participants) | 17
percentage of participants with PFS | 82 [57 to 96]

2. Secondary Outcome: Overall Tumor Response Rate (OR)
Description: To determine overall tumor response rate [% complete response (CR) + % partial response (PR) by RECIST 1.1]. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR) is a disappearance of all target lesions. Partial Response (PR) is a >=30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 17
percentage of participants | 0 [0 to 20]

3. Secondary Outcome: Clinical Benefit Rate
Description: To determine the clinical benefit rate [% CR + % PR + % stable disease by RECIST 1.1] at 6 months. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR) is a disappearance of all target lesions. Partial Response (PR) is a >=30% decrease in the sum of the longest diameter of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 17
percentage of participants | 47 [23 to 72]

ADVERSE EVENTS:
Arm/Group | Nilotinib
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=17)
Fatigue (General disorders) | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=17)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Lung infection (Infections and infestations) | 1
Restlessness (Psychiatric disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Chest pain - cardiac (Cardiac disorders) | 1
Scleral disorder (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 4
Edema face (General disorders) | 1
Fatigue (General disorders) | 8
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 2
Upper respiratory infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 2
Lipase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No